CLINICAL TRIAL: NCT01877512
Title: Effect of Growth Hormone Replacement Therapy on Cardiovascular Risk Factors in Adult Patients With Severe Growth Hormone Deficiency: Association With IGF-I Concentration
Brief Title: GH and Cardiovascular Risk Factors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Prof. dr. M.L. Drent, MD PhD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/12; U1111-1142-9659 (Other: Universal Trial Number); 2012-005066-36 (EudraCT Number)
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Growth Hormone Deficiency; Cardiovascular Diseases; Metabolic Syndrome; Cognition; Physical Activity
MeSH Terms: conditions — Dwarfism, Pituitary; Cardiovascular Diseases; Metabolic Syndrome; Motor Activity

ARMS (2):
- Low dose Growth Hormone (Active Comparator): Halve of the group of men and group of women will receive a decrease of their regular dose of Growth Hormone treatment, with the IGF-I target level of -2 - -1 SD score (low dose=LD).
  Interventions: Drug: Change in daily dosage of Growth Hormone
- High dose Growth Hormone (Active Comparator): Halve of the group of men and group of women will receive an increase of their regular dose of Growth Hormone treatment, with the IGF-I target level of 1 - 2 SD score (high dose=HD).
  Interventions: Drug: Change in daily dosage of Growth Hormone

INTERVENTIONS:
Drug: Change in daily dosage of Growth Hormone
  Other Names: Change in daily dosage of Somatropin

SUMMARY:
Rationale: Abnormally low and high levels of insulin-like growth factor-I (IGF-I) are both associated with increased metabolic risk. Since (U-shaped) associations of IGF-I, within the normal range, have also been found with cardiovascular risk factors and disease in the general population, it would be interesting to investigate if this association can also be found in growth hormone deficient (GHD) adults treated with Growth Hormone (GH). This could be of interest for endocrinologists prescribing GH in clinical practice because strict dosing may become even more important. Next to that, scientific evidence for clinical practice is wanted.

Objective: Next to cardiovascular risk factors (main objectives: body composition and lipid profile; secondary objectives: remainder) we investigate the effect on glucose metabolism, physical performance, and neuropsychological functioning of different levels of IGF-I in GH treated GHD men and women.

Study design: Open-label randomized trial.

Study population: At least 32 subjects, both childhood as adult onset GHD men and women, receiving GH treatment for at least one year, with an age between 20 and 65 years.

Intervention: At entry subjects are already receiving GH treatment according to general clinical practice, and are expected to demonstrate an IGF-I concentration of 0 - 1 SD score (SDS) (normal dose). The group of men and group of women will be randomized to receive either a decrease of their regular dose of GH treatment (IGF-I target level of -2 - -1 SDS) (low dose), or an increase of their regular dose, (IGF-I target level of 1 - 2 SDS) (high dose) for at least 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing surveillance at our centre (VUmc)
* Stable substitution therapy for other pituitary hormone deficiencies

Exclusion Criteria:

* Subjects with a craniopharyngioma as cause of their GHD or pituitary deficiencies
* Contraindications for the use of GH treatment
* (Receiving treatment for) malignant disease (in the past)
* Cardiovascular event less than one year prior to inclusion
* Participation in other studies
* Subjects, who in the opinion of the investigator, are unsuitable in any other way to participate in this study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in cardiovascular risk (body composition and lipid profile) | 24 weeks

SECONDARY OUTCOMES:
Change in cardiovascular risk (inflammatory markers, vascular stiffness, endothelial function, presence of the metabolic syndrome) | 24 weeks
Change in physical performance (muscle strength, physical activity) | 24 weeks
Change in glucose metabolism (fasting and 2hr postprandial glucose, insulin resistance) | 24 weeks
Change in neuropsychological functioning (QoL, cognition, mood) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine L. Drent, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, PO Box 7057, Netherlands

REFERENCES:
- [Derived] van Bunderen CC, Meijer RI, Lips P, Kramer MH, Serne EH, Drent ML. Titrating Growth Hormone Dose to High-Normal IGF-1 Levels Has Beneficial Effects on Body Fat Distribution and Microcirculatory Function Despite Causing Insulin Resistance. Front Endocrinol (Lausanne). 2021 Feb 9;11:619173. doi: 10.3389/fendo.2020.619173. eCollection 2020. PMID 33633687
- [Derived] van Bunderen CC, Deijen JB, Drent ML. Effect of low-normal and high-normal IGF-1 levels on memory and wellbeing during growth hormone replacement therapy: a randomized clinical trial in adult growth hormone deficiency. Health Qual Life Outcomes. 2018 Jul 6;16(1):135. doi: 10.1186/s12955-018-0963-2. PMID 29980224